CLINICAL TRIAL: NCT01520077
Title: A Pilot Study To Evaluate the Efficacy of Vytorin (Simvastatin +Ezetimibe) In the Treatment of Alopecia Areata
Brief Title: Vytorin in the Treatment of Alopecia Areata
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Schachner, Chairman of department of Dermatology & Cutaneous Surgery, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eprost-20100451
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Alopecia Areata
Keywords: alopecia areata; vytorin; statin; hair growth
MeSH Terms: conditions — Alopecia Areata | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vytorin (Other): Subjects will receive Vytorin for 24 weeks. At 24 weeks if regrowth greater or equal than 20%, subjects will be randomized 1/1 to either stop or continue vytorin. Subjects will be follow for additional 24 weeks.
  Subjects that at 24 weeks don't meet the 20% regrowth will be dropped out of the study.
  Interventions: Drug: vytorin

INTERVENTIONS:
Drug: vytorin — Patient will take once per day by mouth Vytorin 10/40mg. Will take it for 24 weeks and then continue or discontinue treatment at that time and be monitored for 24 more weeks. Should there be no improvement by the initial 24 weeks then they will no longer be in the study.
  Other Names: Vytorin 10/40

SUMMARY:
Subjects, non pregnant/lactating and over 18years old, with 40% alopecia areata will take vytorin (statin/ezetimibe) for 24 or 52 weeks and be monitored for hair regrowth.

The investigators hypothesize that Vytorin medication may have an effect on the inflammatory process of alopecia areata. Inactivating the inflammatory process may help in permitting hair regrowth in those subjects.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the efficacy of oral simvastatin + ezetimibe (Vytorin) in treating alopecia areata in subjects 18 years and older.

Secondary objective:

To investigate the presence of heat shock proteins in alopecia areata subjects, before and after treatment with oral simvastatin.

Subjects will be asked to take vytorin 10/40 for a period of 24 or 52 weeks and monitored for progression of hair regrowth. They will have Lipids, creatinine kinase (CK), liver function tests (LFTs), obtained on baseline visit prior to starting the medication and at visit 2, week 8. LFTs will be continuously monitored at visit 4, 7, week 24 and week 40.

In case of muscular pain or tenderness the medication will be stopped immediately. In most cases, muscle symptoms and CK increases resolved when simvastatin treatment was promptly discontinued.

All adverse events will be recorded

The investigators are going to exclude:

oChildren less than 18 years

* Pregnant women
* Lactating women
* Subjects with kidney, liver or muscle disease
* Allergy to the drug or its components. Subjects with history of uncontrolled hypothyroidism, The investigators Hypothesize that this medication may have an effect on the inflammatory process of alopecia areata. Inactivating the inflammatory cascade may help in permitting hair regrowth in those subjects.

ELIGIBILITY:
Inclusion Criteria:

* 40-80% hair loss.
* Clinical diagnosis of alopecia areata
* 18-years or older

Exclusion Criteria:

1. You are less than 18 years old
2. You are pregnant or planning to be pregnant during the next 12 months.
3. You are nursing a child.
4. You have kidney, liver or muscle disease.
5. You have an allergy to Lidocaine, the study drug or its components.
6. You are presently participating in another clinical trial
7. You are currently using, or have used within the past 3 months, the following:

   * Systemic corticosteroids. (prednisone, methylprednisolone, hydrocortisone etc.)
   * Immunosuppressant agents.(cyclosporine, efalizumab etc.)
   * Any medication that may have interaction with Vytorin (check with the study doctor for other medications you are taking).
8. You are currently using, or have used within the past 2 weeks, any topical medication for the treatment of alopecia areata
9. You have an ongoing hypothyroid problem that is not being treated. If this problem is being treated then you can participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
20% Hair regrowth | 6 months
  would like at least 20% regrowth within 6 months time.

SECONDARY OUTCOMES:
maintenance of hair | 6 months
  Will monitor patients from week 25-52 who have had 20% hairgrowth by week 24 and determine if without the medication if they continue to have hairgrowth, remain stable or lose hair.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Schachner, M.D, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Ali A, Martin JM 4th. Hair growth in patients alopecia areata totalis after treatment with simvastatin and ezetimibe. J Drugs Dermatol. 2010 Jan;9(1):62-4. PMID 20120427